CLINICAL TRIAL: NCT01762969
Title: Modification of Imatinib to Other Tyrosine Kinase Inhibitors Dependent on 3-months Molecular Response of CML Patients
Brief Title: Treatment Modification Based on Early Assessment of CML Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Rambam Health Care Campus (Other); Wolfson Medical Center (Other Government); Bnai Zion Medical Center (Other Government); HaEmek Medical Center, Israel (Other); Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, LIAT VIDAL FISHER, Dr., Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML-IS001
Record Dates: First submitted 2013-01-06; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: CML

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modified by molecular response (Experimental): Patients will be treated with imatinib upon diagnosis of CML. Molecular response will be assessed at 3 months of therapy. Based on molecular response imatinib will be continued or changed to another TKI
  Interventions: Other: Treatment modification based on molecular response at 3 months

INTERVENTIONS:
Other: Treatment modification based on molecular response at 3 months — Patients will be treated with imatinib upon diagnosis of CML. Molecular response will be assessed at 3 months of therapy. Based on molecular response imatinib will be continued or changed to another TKI

SUMMARY:
The investigators will check the feasibility of using early molecular response for making treatment decisions. Patients diagnosed with chronic myeloid leukemia will commence imatinib treatment. After 3 months of treatment their response will be assessed. If molecular response would be less the 10% (BCR-ABL1/ABL ISI >10%)imatinib therapy will be stopped and patients will start a different TKI (as nilotinib, dasatinib). The investigators will follow on lab and clinical outcomes.

DETAILED DESCRIPTION:
Objectives:

To establish a national protocol for the treatment of patients with CML. Patients will be stratified by molecular response, and treatment will be adjusted accordingly.

Secondary outcomes To compare clinical outcomes of patients at high risk (transcript level above 10%) to those at low risk (<10%) while using the early switch approach To evaluate the prognostic value of EUTOS, HASFORD, and SOKAL scores using the early switch strategy Patients Patients may be enrolled to the protocol prior to any TKI treatment or at any time point from commencement of imatinib (started at 400 mg daily) and prior to 3 months assessment, if all the necessary baseline data is available, and all other inclusion criteria are met (patients will be excluded if they received treatment with a tyrosine kinase inhibitor other than imatinib)

Inclusion criteria:

1. Adult patients within 6 months after the diagnosis of Philadelphia chromosome-positive CML in the chronic phase

   1. who were not previously treated (with the exception of hydroyurea) for CML or
   2. who were treated with imatinib for CML for up to 3 months, and prior to 3 months assessment (patients will be excluded if they received treatment with a tyrosine kinase inhibitor other than imatinib).
2. Age > 18 years Diagnosis of CML will be made by conventional cytogenetic (chromosome banding analysis) and/or interphase fluorescent in situ hybridization (FISH) analysis of bone marrow containing at least one Philadelphia chromosome-positive metaphase cell. If BCR-ABL1 fusion gene (Philadelphia chromosome) is not detected by conventional cytogenetic analysis, the diagnosis of CML can be confirmed based on FISH analysis or molecular analysis (demonstration of bcr-abl by polymerase chain reaction (PCR)).

Inclusion of patients with any organ dysfunction (cardiac, renal, respiratory, liver) can be done based on the decision of the treating physician.

Exclusion criteria:

Patients will be excluded if they received treatment with a tyrosine kinase inhibitor other than imatinib (i.e., nilotinib, dasatinib) before study entry. Patients may take hydroxyurea or anagrelide for up to 4 weeks prior to imatinib treatment.

Interventions Imatinib 400 mg once daily Response will be assessed after 3 months of therapy. A complete blood count to assess hematologic response and a bone marrow biopsy and/or aspirate, including cytogenetic analysis and molecular analysis for quantitative RT-PCR for BCR-ABL1/ABL will be performed.

Response assessment Assessment of response by molecular analysis of bcr-abl1 will be performed in certified and standardized laboratories (a list of certified laboratories will be distributed).

If a patients has achieved CHR and BCR-ABL1/ABL ISI <10% at 3 months then imatinib will be continued at the dose of 400 mg daily.

If a patient has achieved CHR and BCR-ABL1/ABL ISI >10% at 3 months then imatinib will be stopped and nilotinib 300 mg twice daily or dasatinib 100 mg once daily will be instituted. ECG will be done prior to any change of therapy.

Mutation analysis is recommended prior to the commencement of nilotinib or dasatinib.

Patients will continue to receive the study treatment until the disease will progress or unacceptable toxic effects will developed. In the event of disease progression or the occurrence of adverse event treatment can be stopped or changed under the discretion of the treating physician.

Outcomes Rate of CCyR at 12 months CCyR is defined as absence of Ph-positive metaphases, determined on the basis of G-banding in at least 20 cells in metaphase per bone marrow sample Overall survival Rate of major molecular response at 6, 12, 18, 24 months Cumulative rate of optimal response at 12, 18 months

PFS:

Time from commencement of imatinib till meeting ELN criteria for failure, progression to AP/BC, or death from any cause

EFS:

Time from commencement of imatinib till meeting ELN criteria for failure, progression to AP/BC, grade 3 to 4 adverse event, drug discontinuation (except of the change of imatinib at 3 months according to molecular response), or death from any cause

Safety:

Adverse events will be classified according to the CTCAE NCI US v.3.0 Severe AE

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients within 6 months after the diagnosis of Philadelphia chromosome-positive CML in the chronic phase

  1. who were not previously treated (with the exception of hydroyurea) for CML or
  2. who were treated with imatinib for CML for up to 3 months, and prior to 3 months assessment (patients will be excluded if they received treatment with a tyrosine kinase inhibitor other than imatinib).

     2. Age > 18 years Diagnosis of CML will be made by conventional cytogenetic (chromosome banding analysis) and/or interphase fluorescent in situ hybridization (FISH) analysis of bone marrow containing at least one Philadelphia chromosome-positive metaphase cell. If BCR-ABL1 fusion gene (Philadelphia chromosome) is not detected by conventional cytogenetic analysis, the diagnosis of CML can be confirmed based on FISH analysis or molecular analysis (demonstration of bcr-abl by polymerase chain reaction (PCR)).

     Inclusion of patients with any organ dysfunction (cardiac, renal, respiratory, liver) can be done based on the decision of the treating physician.

     Exclusion Criteria:

     Patients will be excluded if they received treatment with a tyrosine kinase inhibitor other than imatinib (i.e., nilotinib, dasatinib) before study entry. Patients may take hydroxyurea or anagrelide for up to 4 weeks prior to imatinib treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete cytogenetic response | 12 months

SECONDARY OUTCOMES:
Overall survival | 12 months
Rate of major molecular response | 12, 24 months
  Cumulative rate of optimal response at 12, 18 months
PFS | 12 months
  Time from commencement of imatinib till meeting ELN criteria for failure, progression to AP/BC, or death from any cause
Severe Adverse events | 12 months
  Adverse events will be classified according to the CTCAE NCI US v.3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel